CLINICAL TRIAL: NCT07294638
Title: A Humanized Ferritin-Based NIR Fluorescent Probe for Discrimination Between Benign and Malignant Sentinel Lymph Nodes in Early Gastric Cancer
Brief Title: Novel Humanized Ferritin-Based NIR Fluorescent Probe for Identifying Sentinel Lymph Node Metastasis in Early Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-326
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Molecular Imaging
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Humanized Ferritin Probe - Indocyanine green (VE/CX-FTn-ICG): Freshly resected gastric cancer specimens were injected ex vivo via the submucosal layer with the targeted probe VE/CX-FTn-ICG solution for about 60 minutes, followed by fluorescence imaging using a DPM system. The results were analyzed to identify metastatic lymph nodes within the sentinel lymph nodes.
  Interventions: Diagnostic Test: VE/CX-FTn-ICG injection solution

INTERVENTIONS:
Diagnostic Test: VE/CX-FTn-ICG injection solution — The freshly resected gastric cancer specimens were submucosally injection with VE/CX-FTn-ICG solution and underwent fluorescence imaging.

SUMMARY:
With the widespread adoption of early cancer screening, the proportion of early gastric cancer (EGC) in China has been gradually increasing. The primary treatments for EGC are endoscopic and surgical interventions. For EGC invading the submucosal layer, the lymph node metastasis rate is approximately 20%. In clinical practice, subtotal gastrectomy combined with D2 lymphadenectomy is commonly performed to achieve radical tumor resection, resulting in up to 80% of patients undergoing unnecessary lymph node dissection. Sentinel lymph nodes (SLNs), which are the first potential sites along the lymphatic drainage pathway from the primary tumor to receive cancer cells, can effectively represent the status of lymphatic metastasis. As gastric cancer surgery evolves toward minimally invasive, precise, and individualized approaches, there is an urgent clinical need for a safe and effective SLN mapping technique to intraoperatively distinguish between benign and malignant SLNs, thereby avoiding unnecessary lymphadenectomy and improving patient prognosis.

Currently, indocyanine green (ICG) is the only clinically approved near-infrared (NIR) fluorescent dye and is relatively widely used. However, it lacks targeting specificity, diffuses too rapidly, and has difficulty identifying micrometastases in SLNs. Therefore, we aimed to enhance ICG's targeting ability toward metastatic tumor cells to increase fluorescence signal intensity in malignant SLNs, enabling intraoperative differentiation between benign and malignant SLNs and reducing unnecessary lymph node dissection. Considering the high heterogeneity of tumor cells and the molecular diversity among metastatic foci within malignant SLNs, our team innovatively proposed a multi-target probe design to improve targeting capability against heterogeneous tumor cells. Based on molecular imaging technology combined with near-infrared (NIR) imaging, we developed a humanized ferritin-based probe (VE/CX-FTn) targeting metastatic lymph nodes. Previous studies have confirmed the effective identification of metastatic lymph nodes by the VE/CX-FTn probe.

To further validate the effectiveness of this probe in identifying SLN metastasis in early gastric cancer with a low lymph node metastasis rate, this study plans to use residual early gastric cancer tissues obtained from post-surgical resections to evaluate the probe's imaging capability for SLNs. Furthermore, a prospective clinical sample cohort study will be conducted to verify its diagnostic efficacy for metastatic lymph nodes of varying sizes. The aim is to demonstrate that our developed probe can guide the identification of SLNs in early gastric cancer and assist in determining the presence of SLN metastasis, thereby reducing unnecessary lymphadenectomy and improving patient prognosis.

This study employs a novel NIR fluorescent molecular probe, VE/CX-FTn-ICG, based on humanized ferritin, with the objective of investigating its effectiveness in distinguishing between benign and malignant sentinel lymph nodes in early gastric cancer. Using this probe, we have already demonstrated that VE/CX-FTn-ICG enables precise differentiation between benign and malignant lymph nodes in animal models. The probe specifically binds to tumor cells, exhibiting high targeting specificity and imaging capability, thereby providing real-time and accurate intraoperative imaging of SLNs for early gastric cancer surgery. A further goal of this study is to validate the application efficacy of this targeted probe in distinguishing between benign and malignant SLNs using ex vivo human early gastric cancer tissue samples. This aims to provide a reliable auxiliary tool for intraoperative SLN biopsy in early gastric cancer, assisting in avoiding unnecessary lymph node resection for patients, and ultimately improving surgical outcomes and patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed early gastric cancer eligible for radical resection, with histologically verified adenocarcinoma component (cT1-cT2, tumor diameter ≤4 cm);Age≥18years；No gender restriction；voluntary participation with written informed consent.

Exclusion Criteria:

* Patients deemed ineligible for participation by the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was recruited from the Nanfang Hospital of Southern Medical University in Guangzhou, China.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
1. The area under the curve (AUC) value of the humanized targeted probe (VE/CX-FTn-ICG) for diagnosing sentinel lymph node metastasis in early gastric cancer | 1 year
1. The area under the curve (AUC) value of the humanized targeted probe (VE/CX-FTn-ICG) for diagnosing sentinel lymph node metastasis in early gastric cancer | 1 years
  Pathologists performed histopathological examination of the sentinel lymph nodes，while researchers compared the SLNs identified by pathological results with those predicted by the fluorescence imaging of the probe to calculate the AUC value of VE/CX-FTn-ICG.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University , Guangzhou, Guangzhou, Guangdong, China